CLINICAL TRIAL: NCT01645566
Title: Impact of a Task Focusing Strategy on Perceived Stress Levels and Performance During a Simulated Cardiopulmonary Resuscitation: A Randomized Controlled Trial
Brief Title: Task Focusing Strategy During a Simulated Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Philipp Schuetz, Dr., University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BS1330978
Record Dates: First submitted 2012-07-15; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Mental Stress
Keywords: cardiopulmonary resuscitation; stress; intervention
MeSH Terms: conditions — Stress, Psychological | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): instructions about focusing on relevant task elements by posing two task-focusing questions ("what is the patient's condition?", "what immediate action is needed?") when feeling overwhelmed by stress (intervention-group)
  Interventions: Behavioral: instruction
- Control (No Intervention): No instructions

INTERVENTIONS:
Behavioral: instruction — instructions about focusing on relevant task elements by posing two task-focusing questions ("what is the patient's condition?", "what immediate action is needed?") when feeling overwhelmed by stress (intervention-group)
  Arms: intervention

SUMMARY:
This is a prospective randomized controlled study. The aim of this study is to

1. describe the stress patterns experienced during a CPR situation;
2. investigate whether the perceived stress was associated with CPR performance in terms of hands-on time and time to start CPR;
3. to investigate whether this task focusing strategy reduces perceived stress levels, and
4. whether this translates into better CPR performance. Based on findings that clear, directive leadership can enhance performance in cardiac resuscitation, we further 5) investigate if stress was associated with fewer leadership statements.

ELIGIBILITY:
Inclusion Criteria:

* 4th year medical students

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
perceived levels of stress and feeling overwhelmed (stress/overload) | time from start of CPR until scenario is finished (usually 5-10min)
  This is a simulator study and the study starts after students entered the simulator and the manikin has a cardiac arrest. The scenarios usually last for not more than 5-10 min at which time point the study is finished

SECONDARY OUTCOMES:
hands-on time | time from start of CPR until scenario is finished (usually 5-10min)
  This is a simulator study and the study starts after students entered the simulator and the manikin has a cardiac arrest. The scenarios usually last for not more than 5-10 min at which time point the study is finished
time to start CPR | time from start of CPR until scenario is finished (usually 5-10min)
Number of leadership statements | time from start of CPR until scenario is finished (usually 5-10min)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hunziker, MD, MPH, Principal Investigator — University Hospital Basel, Medical Intensive Care Unit
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Hunziker S, Semmer NK, Tschan F, Schuetz P, Mueller B, Marsch S. Dynamics and association of different acute stress markers with performance during a simulated resuscitation. Resuscitation. 2012 May;83(5):572-8. doi: 10.1016/j.resuscitation.2011.11.013. Epub 2011 Nov 22. PMID 22115935
- [Background] Hunziker S, Laschinger L, Portmann-Schwarz S, Semmer NK, Tschan F, Marsch S. Perceived stress and team performance during a simulated resuscitation. Intensive Care Med. 2011 Sep;37(9):1473-9. doi: 10.1007/s00134-011-2277-2. Epub 2011 Jun 22. PMID 21695475
- [Background] Hunziker S, Johansson AC, Tschan F, Semmer NK, Rock L, Howell MD, Marsch S. Teamwork and leadership in cardiopulmonary resuscitation. J Am Coll Cardiol. 2011 Jun 14;57(24):2381-8. doi: 10.1016/j.jacc.2011.03.017. PMID 21658557
- [Derived] Hunziker S, Pagani S, Fasler K, Tschan F, Semmer NK, Marsch S. Impact of a stress coping strategy on perceived stress levels and performance during a simulated cardiopulmonary resuscitation: a randomized controlled trial. BMC Emerg Med. 2013 Apr 22;13:8. doi: 10.1186/1471-227X-13-8. PMID 23607331